CLINICAL TRIAL: NCT06035198
Title: Developement of Prognosis Predictive Precision Medicine Based on a Digital Twin Reflecting the Motor Patterns in Stroke Patients
Brief Title: Developement of Stroke Prognosis Predictive Precision Medicine Based on a Digital Twin
Status: Recruiting | Type: Observational
Sponsor: Seyoung Shin (Other)
Responsible Party: Sponsor-Investigator, Seyoung Shin, Principal Investigator, CHA University
Organization: CHA University (Other)
Other Study IDs: RS-2023-00262005
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Patients diagnosed with stroke at four hospitals in Korea
  Interventions: Other: Stroke

INTERVENTIONS:
Other: Stroke — No intervention

SUMMARY:
The purpose of this study is to realize customized precision medicine for stroke patients and the visual digitization of patient medical information required in the era of digital transformation.

This study will collect large-scale, high-quality clinical data and daily life exercise pattern data covering the subacute to chronic stages of stroke patients. Based on this, we will use artificial intelligence analysis technology to predict the functional status of stroke patients in the chronic stage after their disability is fixed. We aim to develop the next generation of personalized digital twins by creating a prognostic prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years of age with a history of stroke onset between 2018.01.01 to 2023.07.31.
* Patients who exist rehabilitation medical evaluation after stroke onset
* Patients who voluntarily decide to participate in this study

Exclusion Criteria:

* Those who have severe internal diseases such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc. and are in poor overall condition.
* Those who have impaired ability to consent (MMSE score less than 10 points) and not accompanied by a care-giver.
* In any other cases where the researcher determines that participation in this study is not appropriate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients receiving treatment at four hospitals in Korea
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Barthel Index (MBI) | minimum 6 months to maximum 6 years
  A scale to measure disability or dependence in activities of daily living (ADL) of stroke survivors (range 0-100)

SECONDARY OUTCOMES:
Mini Mental Status Examination (MMSE) | minimum 6 months to maximum 6 years
  Mini-Mental State Examination (MMSE) is a 30-question assessment of cognitive function that evaluates attention and orientation, memory, registration, recall, calculation, language and ability to draw a complex polygon (range 0-30)
Functional Ambulatory Category (FAC) | minimum 6 months to maximum 6 years
  The Functional Ambulation Categories (FAC) is a 6-point functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. (range 0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Seyoung Shin, MD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Gyeonggi-do, South Korea